CLINICAL TRIAL: NCT05226936
Title: Study for Detection of Donor-derived Cell-free DNA After Renal Transplantation Using Devysers NGS-based Chimerism Assay.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Dan Hauzenberger M.D., Ph.D. Assoc. Professor, Karolinska University Hospital Sweden (Unknown)
Responsible Party: Principal Investigator, Prof. Eytan Mor, Director Kidney Transplant Center, Sheba Medical Center
Other Study IDs: 9024-21-SMC
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Cell-Free Nucleic Acids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood serum and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cell free DNA analysis — samples will be analysed using molecular techniques including sequencing for measuring dd-cfDNA or analysis of the presence of HLA-antibodies using commercial bead-technologies (Luminex or Immucor)
  Other Names: Donor Specific Antibody analysis

SUMMARY:
The aim of this study is to evaluate highly sensitive quantitative tests for early molecular detection of graft rejection and associated immune response from liquid biopsies in the blood from patients undergoing renal transplantation and secondly, to evaluate the evolution of de-novo HLA antibodies following renal transplantation. Furthermore, we are interested in the correlation of tissue damage caused by rejection, as measured by the presence of dd-cfDNA, and the presence of de-novo HLA antibodies.

DETAILED DESCRIPTION:
Each year 40-60 patients undergo renal transplant with a living donor (LD) at Karolinska University Hospital. Prior to transplantation, these patients and their donors are investigated for their immunological compatibility. This includes cytotoxic- and flow cytometric crossmatches, HLA typing as well as determination of possible presence of panel-reactive HLA antibodies (PRA). Normally these investigations are performed 2-3 months prior to renal transplantation. Once a patient has been accepted for transplantation with a given living donor, they will, prior to transplantation be asked whether they are interested in taking part of the present study. If the patient and the donor do accept, we will collect 15 mL of blood prior to transplantation using suitable sample collection tubes (Cell-Free BCT tubes). This sample will be used for screening patient and donor for specific genetic markers. Furthermore, the pretransplant samples will be used for determining the presence or absence of HLA antibodies for each patient. We aim to include up to 50 patients in the current study.

During the first 24-48 hrs after transplantation, two more samples (10 mL) from the patient will be collected to measure the potential presence of dd-cfDNA including cell-free particles such as exosomes. The cell-free DNA and RNA from all samples will be extracted, stored frozen and later sequenced. Following transplantation and initiation of the immunosuppressive therapy, samples for analysis will be obtained once every week for up to 3 months. All collected samples will be either analysed immediately or frozen for future analysis. Stored frozen samples could, at a later time point, be thawed, batched and analysed using molecular techniques including sequencing for measuring dd-cfDNA or analysis of the presence of HLA-antibodies using commercial bead-technologies (Luminex or Immucor). Results from these assays will be added to a dedicated database. The obtained laboratory results will be compared to clinical outcome including graft survival, patient survival, clinical and subclinical rejections etc. as well as other laboratory data (e.g. results from pathological examination of the graft, clinical chemistry, concentration of immunosuppressive drugs etc).

ELIGIBILITY:
Inclusion Criteria:

Patients older than 20 undergoing kidney transplantation -

Exclusion Criteria:

Patients included in other studies Patients a combined transplant with other donor Patients not eligible to sign an inform consent Patients with primary non-function or those that lost their graft during the first 3 months

-

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing live donor or deceased donor transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Degree of chimerism | According to the study protocol before and after transplantation in defined intervals up to 3 moths
  The fraction of cell free donor DNA will be measured after transplant

IPD SHARING:
Plan to Share IPD: Yes
The study is in collaboration with the transplant center in Sweden. Each study patients will be given a code and the coded information will be shared with our partners
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: The data will be available for 3 yeras from the completion of the recuitment of all patients
Access Criteria: Shared mail with an access code

REFERENCES:
- [Background] Bloom RD, Bromberg JS, Poggio ED, Bunnapradist S, Langone AJ, Sood P, Matas AJ, Mehta S, Mannon RB, Sharfuddin A, Fischbach B, Narayanan M, Jordan SC, Cohen D, Weir MR, Hiller D, Prasad P, Woodward RN, Grskovic M, Sninsky JJ, Yee JP, Brennan DC; Circulating Donor-Derived Cell-Free DNA in Blood for Diagnosing Active Rejection in Kidney Transplant Recipients (DART) Study Investigators. Cell-Free DNA and Active Rejection in Kidney Allografts. J Am Soc Nephrol. 2017 Jul;28(7):2221-2232. doi: 10.1681/ASN.2016091034. Epub 2017 Mar 9. PMID 28280140
- [Background] Everly MJ, Terasaki PI. Monitoring and treating posttransplant human leukocyte antigen antibodies. Hum Immunol. 2009 Aug;70(8):655-9. doi: 10.1016/j.humimm.2009.04.019. Epub 2009 Apr 15. PMID 19375466
- [Background] Lee PC, Zhu L, Terasaki PI, Everly MJ. HLA-specific antibodies developed in the first year posttransplant are predictive of chronic rejection and renal graft loss. Transplantation. 2009 Aug 27;88(4):568-74. doi: 10.1097/TP.0b013e3181b11b72. PMID 19696641